CLINICAL TRIAL: NCT02735512
Title: MDSC Clinical Assay for Cancer Detection and Monitoring in Bladder Carcinoma
Brief Title: MDSC Clinical Assay in Finding and Monitoring Cancer Cells in Blood and Urine Samples From Patients With or Without Localized or Metastatic Bladder Cancer
Status: Terminated | Type: Observational
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4B-15-2; NCI-2016-00265 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4B-15-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-03-15; First posted 2016-04-12 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: No Evidence of Disease; Stage II Bladder Cancer; Stage III Bladder Cancer; Stage IVA Bladder Cancer; Stage IVB Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: Patients without cancer undergo collection of blood and urine samples for analysis via MDSC clinical assay at baseline, 1 week, and 4 months.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Group II: Patients with localized bladder cancer undergo collection of blood and urine samples for analysis via MDSC clinical assay at baseline, 1 week, and within 4 weeks after cystectomy.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis
- Group III: Patients with metastatic cancer undergo collection of blood and urine samples for analysis via MDSC clinical assay at baseline, 1 week, and within 4 weeks after completion of 4 courses of systemic chemotherapy.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of blood and urine samples
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Samples undergo MDSC clinical assay

SUMMARY:
This pilot research trial studies how well myeloid derived suppressor cells (MDSC) clinical assay works in finding and monitoring cancer cells in blood and urine samples from patients with or without localized or metastatic bladder cancer. Studying samples of blood and urine from patients with or without bladder cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer and may help doctors improve ways to diagnose and treat patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate a novel clinical assay (MDSC clinical assay) to detect cancer associated immune cells in the peripheral blood of patients as a means to better detect and monitor malignant bladder cancer in patients.

II. Estimate mean MDSC level, intra-patient variability, and inter-patient variability, for 3 groups of subjects with variable bladder cancer disease status at baseline.

III. In patients with known localized, muscle-invasive bladder cancer who undergo surgical treatment: to determine the change in MDSC level from baseline to after treatment including surgery.

IV. In patients with known metastatic bladder cancer who undergo systemic treatment: to determine the change in MDSC level from baseline to after 4 cycles of treatment compared to the change in tumor burden as evaluated by radiographic imaging.

V. In patients with no history of cancer: to determine the changes in MDSC levels from baseline to after 4 months.

SECONDARY OBJECTIVES:

I. Compare MDSC level measurements to urine cytology analysis at baseline and after treatment to determine whether the two tests correlate in any of the 3 groups of patients defined in this study.

OUTLINE:

GROUP I: Patients without cancer undergo collection of blood and urine samples for analysis via MDSC clinical assay at baseline, 1 week, and 4 months.

GROUP II: Patients with localized bladder cancer undergo collection of blood and urine samples for analysis via MDSC clinical assay at baseline, 1 week, and within 4 weeks after cystectomy.

GROUP III: Patients with metastatic cancer undergo collection of blood and urine samples for analysis via MDSC clinical assay at baseline, 1 week, and within 4 weeks after completion of 4 courses of systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the criteria for one of the three following groups:

  * Normal patients- aged 40 years and older with no evidence of hematuria or cancer
  * Patients with localized bladder cancer diagnosed by cystoscopy and pathology: T2N0M0 or T3N0M0 who have not received neoadjuvant chemotherapy
  * Patients with metastatic bladder cancer: newly diagnosed with no previous treatment for metastatic disease
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* For normal subject arm: evidence of cancer or hematuria
* For localized bladder cancer: evidence of metastatic disease, second cancer, prior chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* For metastatic bladder cancer: prior therapy for metastatic disease
* Uncontrolled intercurrent illness including, but not limited to previous or current history of second malignancy unrelated to bladder cancer; autoimmune disease or immune deficiency, chronic treatment with immunomodulatory therapies (e.g. glucocorticoids); significant trauma, surgery, or infection in the past two weeks or psychiatric illness/social situations that would limit compliance with study requirements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal patients- aged 40 years and older with no evidence of hematuria or cancer Patients with localized bladder cancer diagnosed by cystoscopy and pathology: T2N0M0 or T3N0M0 who have not received neoadjuvant chemotherapy Patients with metastatic bladder cancer: newly diagnosed with no previous treatment for metastatic disease
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Change in MDSC level in patients with known localized, muscle-invasive bladder cancer who undergo surgical treatment | Baseline to up to 4 months
Change in MDSC level in patients with known metastatic bladder cancer who undergo systemic treatment | Baseline to up to 6 months
  The direction and magnitude of the changes in Group 3 will be compared to the changes in tumor burden assessed radiographically - to explore the associations.
Change in MDSC level in patients with no history of cancer | Baseline to 4 months
Change in tumor burden evaluated by radiographic imaging | Baseline to up to 1 year

SECONDARY OUTCOMES:
Change in urine cytology analysis | Baseline to up to 4 months
  The MDSC levels at baseline will be compared (plots and correlations) to the urine cytology levels (Groups 2 and 3) to describe any associations; for Group 3, the changes (baseline to post treatment) in the MDSC levels will be compared to the changes in urine cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States